CLINICAL TRIAL: NCT06991985
Title: Analysis of Factors Associated With The Occurrence of Amniotic Fluid Entry in Patients Undergoing Caesarean Section
Acronym: AOFAWTOOAFEIPU
Status: Not yet recruiting | Type: Observational
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Other Study IDs: yuewei20250520
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Amniotic Fluid Embolism
MeSH Terms: conditions — Embolism, Amniotic Fluid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amniotic fluid into the blood group
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay
- the control group
  Interventions: Diagnostic Test: Enzyme-linked immunosorbent assay

INTERVENTIONS:
Diagnostic Test: Enzyme-linked immunosorbent assay — Serum STN and C4 levels were detected

SUMMARY:
To compare serum STN （Neuraminic acid-N-acetylgalactose）antigen concentrations in patients undergoing cesarean section and to study the factors associated with amniotic fluid entry.Compare the serum complement C4 concentration in patients in the amniotic fluid admission group with those in the non-admission group to study whether amniotic fluid admission triggers the body's immune response.To record the patients' blood pressure, heart rate, blood oxygen, and the occurrence of related symptoms and adverse reactions at the time of admission, at the time of blood collection, at the time of discharge from the room, and at the time of the occurrence of haemodynamic changes.

DETAILED DESCRIPTION:
All patients were routinely fasted for 8 h and abstained from drinking for 4 h. After entering the operating theatre, intravenous access was opened, and blood pressure, heart rate, electrocardiogram, oxygen saturation and patient's symptoms were continuously monitored during the operation. After obtaining informed consent for anaesthesia from the patient and his family, intrathecal anaesthesia or general anaesthesia was administered according to the situation. Venous blood was drawn from the patient 30 min after the foetus was dissected out, and samples were preserved to measure the concentration of serum STN antigen and the concentration of complement C4; data were collected through the resident workstation system and the manual anaesthesia system, and the patient's information included age, history of allergy, number of deliveries, and history of combining with other illnesses; and the pregnancy information included Placenta type, amniotic fluid, hypertensive disorders of pregnancy, and whether or not the pregnancy was multiple; delivery data included whether or not elective caesarean section was performed, operator factors, intensity of contractions, method of rupture of membranes, and anaesthesia method.

ELIGIBILITY:
Inclusion Criteria:

* Approved consent and informed consent of the patient by the Ethics Committee of the Second Hospital of Shanxi Medical University;
* ASA classification of I-III;
* Age 20-50 years old;
* No previous history of psychiatric diseases or psychotropic drugs;

Exclusion Criteria:

* Suffer from diseases of the cardiorespiratory system;
* Those with communication difficulties who were unable to complete the screening questionnaire;

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients in the Second Hospital of Shanxi Medical University from May 2025 to November 2025
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
STN | 24 hours
  Serum STN levels
C4 | 24 hours
  Serum C4 levels

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No